CLINICAL TRIAL: NCT01295580
Title: A Multicenter, Randomized, Double-blind, Parallel, Active-controlled Clinical Trial With Non-inferiority Comparison to Evaluate Efficacy and Safety of Intra-articular Injection of DUROLANE® vs. ARTZ® in Treatment of Knee Osteoarthritis
Brief Title: Comparative Study of Safety and Efficacy of Two Hyaluronic Acids for the Treatment of Knee Osteoarthritis Pain
Acronym: DRAGON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bioventus LLC (Industry)
Collaborators: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TG1018DLN
Record Dates: First submitted 2011-02-11; First posted 2011-02-14 (Estimated); Results first posted 2021-04-09 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-03

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigational product was masked from study staff and participants with the exception of the unblinded treating investigator conducting the intra-articular injections.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

ARMS (2):
- ARTZ sodium hyaluronate (Active Comparator): The comparator product, ARTZ, is manufactured by Seikagaku Corporation, Japan. Subjects randomized to the ARTZ group were administered five weekly intra-articular injections (2.5 ml, NASHA 25 mg). ARTZ is a sterile, viscoelastic nonpyrogenic solution of purified, high molecular weight (620,000-1,170,000 daltons) sodium hyaluronate having a pH of 6.8-7.8. The sodium hyaluronate is extracted from chicken combs.
  Interventions: Device: ARTZ
- DUROLANE hyaluronic acid (Active Comparator): The investigational product was provided in pre-filled syringes containing stabilized non-animal hyaluronic acid (20 mg/mL). Only one injection was given for those subjects randomized to the DUROLANE group, followed by 4 sham injections. DUROLANE is free from products of animal origin and is manufactured by Q-Med AB Corporation.The sham injection procedure was same as the active injection, except that they were subcutaneous and an empty syringe was used.
  Interventions: Device: DUROLANE

INTERVENTIONS:
Device: ARTZ — Hyaluronic acid (five 2.5 mL injections)
  Arms: ARTZ sodium hyaluronate
Device: DUROLANE — Hyaluronic acid stabilized (one 3.0 mL injection + four weekly 0 mL sham injections)
  Arms: DUROLANE hyaluronic acid

SUMMARY:
The purpose of this study is to determine the comparative safety and efficacy of intra-articular injection of hyaluronic acid, obtained from two different sources, in the treatment of osteoarthritic pain of the knee.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double blind, parallel-controlled clinical trial using a non-inferiority comparison to evaluate the efficacy and safety of an intra-articular injection of Durolane® vs Artz® in the treatment of knee osteoarthritis. Subjects will be randomized 1:1 to receive either Durolane or Artz. All subjects will be followed up for 26 weeks from the initial treatment.The screening period is expected to be up to 2 weeks in duration before the baseline visit. Each subject will provide a written informed consent and undergo a qualifying screening. Assessment at screening will include postero-anterior view of standing weight-bearing semi-flexed radiographs of the study knee. The osteoarthritis changes of the study knee will be graded 0,1,2,3 or 4 according to the Kellgren-Lawrence radiographic scoring criteria. Radiographic assessment will be made by an assigned and well trained investigator at each study center. The study knee and contralateral knee will use the Likert WOMAC 5-point scoring for pain assessment.

Physical examination of the knees and vital signs will be performed (this examination will be repeated at end).

ELIGIBILITY:
Inclusion Criteria:

* Subject (female or male) 40-80 years of age, inclusive
* Documented diagnosis of mild to moderate osteoarthritis of the study knee that fulfil the ACR(American College of Rheumatology) criteria
* Radiographic evidence of osteoarthritis in the study knee (Kellgren Lawrence radiographic score is 2 or 3)

Exclusion Criteria:

* Clinically apparent tense effusion of the study knee on examination determined by either a positive bulge sign or positive ballottement of the patella
* Kellgren-Lawrence radiographic score 0, 1 or 4 in the study knee
* Symptomatic osteoarthritis of the contralateral knee or of either hip that is not responsive to acetaminophen/paracetamol and/or requires any protocol prohibited therapies

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2011-01; Primary Completion 2011-08 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jianhao Lin, MD, Principal Investigator — People Hospital of Beijing University No. 11 South Ave., Xizhimen, Beijing
Locations (7):
- China (7):
  - Beijing Frienship Hospital, Beijing
  - Beijing General Military Hospital, Beijing
  - Beijing University #3 Hospital, Beijing
  - Beijing University People's Hospital, Beijing
  - Zhejiang #2 Hospital, Hangzhou
  - Shanghai #6 People's Hospital, Shanghai
  - Shanghai #9 People's Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhang H, Zhang K, Zhang X, Zhu Z, Yan S, Sun T, Guo A, Jones J, Steen RG, Shan B, Zhang J, Lin J. Comparison of two hyaluronic acid formulations for safety and efficacy (CHASE) study in knee osteoarthritis: a multicenter, randomized, double-blind, 26-week non-inferiority trial comparing Durolane to Artz. Arthritis Res Ther. 2015 Mar 10;17(1):51. doi: 10.1186/s13075-015-0557-x. PMID 25889322

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ARTZ | DUROLANE
Started | 174 | 175
Completed | 164 | 167
Not Completed | 10 | 8
Not completed — Protocol Violation | 4 | 2
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Adverse Event | 2 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Other: inconvenience | 1 | 0
Not completed — Other: family objection | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ARTZ | DUROLANE | Total
Number analyzed (Participants) | 174 | 175 | 349
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (8.16) | 60.3 (8.11) | 60.4 (8.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 139 | 132 | 271
  Male | 35 | 43 | 78
Race/Ethnicity, Customized [Number; unit: participants]
  Nationality: Han | 173 | 168 | 341
  Nationality: Other | 1 | 7 | 8
Region of Enrollment [Number; unit: participants]
  China | 174 | 175 | 349

OUTCOME MEASURES:

1. Primary Outcome: WOMAC (Western Ontario and McMaster Osteoarthritis Index) Pain Subscale Change From Baseline
Description: Pain assessment is made of 5 items; each has 5 possible values 0=none, 1=mild, 2=moderate, 3=severe, 4=extreme. The items are summed for a total range of 0 to 20. Therefore, the pain change from baseline range is -20 to 20. A negative change is a reduction in pain from the baseline pain score.
  A mixed-effect repeated measures regression model was used to estimate a least square mean for the entire "Measured Time Frame".
  Change from baseline was the dependent variable. Subject baseline score was a fixed effect covariate. Enrollment site, treatment, visit, and treatment by visit interaction were fixed class effects. Subject was a random effect. A least square mean single point estimate and 95%CI was calculated for the entire "Measured Time Frame" using all data collected at each time point within the "Measured Time Frame".
Time Frame: over 18 weeks (week timepoints 6, 10, 14, and 18)
Population: per protocol: all subjects randomized and treated with no important protocol deviation(s), which were established at a blinded data review meeting. An important deviation is any deviation that has the potential to bias the primary outcome.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | ARTZ | DUROLANE
Number analyzed (Participants) | 158 | 161
units on a scale | -5.87 [-6.23 to -5.52] | -5.97 [-6.32 to -5.61]
Statistical Analysis 1: Comparison: ARTZ vs DUROLANE; Primary Hypothesis: Ho: μDUR[18] - μArtz[18] ≥ +1.6 units Ha: μDUR[18] - μArtz[18] < +1.6 units Power Calculations: Assume the over 18 weeks difference is 0mm, SD 20mm (5 on the Likert scale), 90% power, 2-sided test alpha 5%, and a 8mm non-inferiority margin (1.6 on the Likert scale), the sample size required is 132 subjects per group adjusted to 175 to hold power constant due to loss to follow-up and dropout; Test type: Non-Inferiority or Equivalence — This is a non-inferiority test. The non-inferiority margin of +1.6 units corresponds to an 8% margin on the pain subscale (range 0-20) Alpha inflation was controlled using pre-planned stepwise hypotheses testing (1) WOMAC Pain over 18 weeks then (2) over 26 weeks, (3) WOMAC Physical Function over 18 weeks then (4) over 26 weeks, (5) Subject Global Assessment over 18 weeks then (6) over 26 weeks, (7) WOMAC Knee Stiffness over 18 weeks then (8) over 26 weeks; Alpha inflation due to multiple testing was controlled using preplanned ordered stepwise hypothesis testing first over 18 weeks then over 26 weeks. This section reports the first step WOMAC pain over 18 week pain subscale primary analyses; The second step is to test Durolane WOMAC pain non-inferior to Artz WOMAC pain over 26 weeks; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.58 to 0.39]

2. Secondary Outcome: WOMAC (Western Ontario and McMaster Osteoarthritis Index) Pain Subscale Change From Baseline
Description: as for outcome 1
Time Frame: over 26 weeks (week 6, 10, 14, 18, and 26)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | ARTZ | DUROLANE
Number analyzed (Participants) | 158 | 161
units on a scale | -6.05 [-6.39 to -5.71] | -6.15 [-6.49 to -5.81]
Statistical Analysis 1: Comparison: ARTZ vs DUROLANE; Ho: μDUR[26] - μArtz[26] ≥ +1.6 units Ha: μDUR[26] - μArtz[26] < +1.6 units; Test type: Non-Inferiority or Equivalence — This is a non-inferiority test. The non-inferiority margin of +1.6 units corresponds to an 8% margin on the pain subscale (range 0-20); Alpha inflation due to multiple testing was controlled using preplanned ordered stepwise hypothesis testing first pain over 18 weeks then pain over 26 weeks. This section reports the over 26 week pain subscale results; The third ordered test is Durolane WOMAC physical function subscale non-inferior to Artz WOMAC physical function subscale over 18 weeks; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.56 to 0.37]

3. Secondary Outcome: WOMAC (Western Ontario and McMaster Osteoarthritis Index) Physical Function Subscale Change From Baseline
Description: Physical Function assessment is made of 17 items; each has 5 possible values 0=none, 1=mild, 3=moderate, 4=extreme. The items are summed for a total range of 0 to 68. Therefore, the physical function change from baseline range is -68 to 68. A negative change is an improvement in physical function from the baseline physical function score.
  A mixed-effect repeated measures regression model was used to estimate a least square mean for the entire "Measured Time Frame".
  Change from baseline was the dependent variable. Subject baseline score was a fixed effect covariate. Enrollment site, treatment, visit, and treatment by visit interaction were fixed class effects. Subject was a random effect. A least square mean single point estimate and 95%CI was calculated for the entire "Measured Time Frame" using all data collected at each time point within the "Measured Time Frame".
Time Frame: over 18 weeks (week timepoints 6, 10, 14, and 18)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | ARTZ | DUROLANE
Number analyzed (Participants) | 158 | 161
units on a scale | -12.10 [-12.95 to -11.26] | -12.75 [-13.60 to -11.91]
Statistical Analysis 1: Comparison: ARTZ vs DUROLANE; Ho: μDUR[18] - μArtz[18] ≥ +5.44 units Ha: μDUR[18] - μArtz[18] < +5.44 units; Test type: Non-Inferiority or Equivalence — This is a non-inferiority test. The non-inferiority margin of +5.44 units corresponds to an 8% margin on the physical function subscale (range 0-68); Alpha inflation due to multiple testing was controlled using preplanned ordered stepwise hypothesis testing first over 18 weeks then over 26 weeks. This section reports the over 18 week physical function results; The fourth step is to test Durolane WOMAC physical function non-inferior to Artz physical function over 26 weeks; Mean Difference (Final Values) = -0.65, 95% CI 2-sided [-1.81 to 0.51]

4. Secondary Outcome: WOMAC (Western Ontario and McMaster Osteoarthritis Index) Physical Function Subscale Change From Baseline
Description: as for outcome 3
Time Frame: over 26 weeks (week timepoints 6, 10, 14, 18, and 26)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | ARTZ | DUROLANE
Number analyzed (Participants) | 158 | 161
units on a scale | -12.58 [-13.39 to -11.77] | -13.16 [-13.97 to -12.35]
Statistical Analysis 1: Comparison: ARTZ vs DUROLANE; Ho: μDUR[26] - μArtz[26] ≥ +5.44 units Ha: μDUR[26] - μArtz[26] < +5.44 units; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Alpha inflation due to multiple testing was controlled using preplanned ordered stepwise hypothesis testing first over 18 weeks then over 26 weeks. This section reports the over 26 week physical function subscale results; The fifth step is to test Durolane subject global assessment non-inferior to Artz global assessment over 18 weeks; Mean Difference (Final Values) = -0.58, 95% CI 2-sided [-1.69 to 0.53]

5. Secondary Outcome: Subject Global Assessment Change From Baseline
Description: Subject global assessment is one question "Considering all the ways your knee osteoarthritis affects you, how are you doing today?". It has 11 values 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10 labeled only at the extremes; 0 = very bad and 10 = very good. The change from baseline range is -10 to 10. A positive change is an improvement from the baseline subject global assessment score.
  A mixed-effect repeated measures regression model was used to estimate a least square mean for the entire "Measured Time Frame".
  Change from baseline was the dependent variable. Subject baseline score was a fixed effect covariate. Enrollment site, treatment, visit, and treatment by visit interaction were fixed class effects. Subject was a random effect. A least square mean single point estimate and 95%CI was calculated for the entire "Measured Time Frame" using all data collected at each time point within the "Measured Time Frame".
Time Frame: over 18 weeks (week timepoints 6, 10, 14, and 18)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | ARTZ | DUROLANE
Number analyzed (Participants) | 158 | 161
units on a scale | 2.55 [2.33 to 2.77] | 2.70 [2.48 to 2.92]
Statistical Analysis 1: Comparison: ARTZ vs DUROLANE; Ho: μDUR[18] - μArtz[18] ≤ -0.8 units Ha: μDUR[18] - μArtz[18] > -0.8 units; Test type: Non-Inferiority or Equivalence — This is a non-inferiority test. The non-inferiority margin of -0.8 units corresponds to an 8% margin on the subject global assessment (range 0-10). Note that because the assessment interpretation is reversed as compared to the WOMAC assessments the lower bound of the 95%CI is compared to the -0.8 non-inferiority margin; Alpha inflation due to multiple testing was controlled using preplanned ordered stepwise hypothesis testing first over 18 weeks then over 26 weeks. This section reports the over 18 week subject global assessment results; The sixth step is to test Durolane subject global assessment non-inferior to Artz subject global assessment over 26 weeks; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [-0.15 to 0.45]

6. Secondary Outcome: Subject Global Assessment Change From Baseline
Description: as for outcome 5
Time Frame: over 26 weeks (week timepoints 6, 10, 14, 18, and 26)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | ARTZ | DUROLANE
Number analyzed (Participants) | 158 | 161
units on a scale | 2.67 [2.45 to 2.88] | 2.81 [2.59 to 3.02]
Statistical Analysis 1: Comparison: ARTZ vs DUROLANE; Ho: μDUR[18] - μArtz[18] ≤ -0.8 units Ha: μDUR[18] - μArtz[18] > -0.8 units; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Alpha inflation due to multiple testing was controlled using preplanned ordered stepwise hypothesis testing first over 18 weeks then over 26 weeks. This section reports the over 26 week subject global assessment results; The seventh step is to test Durolane WOMAC knee stiffness non-inferior to Artz WOMAC knee stiffness over 18 weeks; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-0.16 to 0.43]

7. Secondary Outcome: WOMAC (Western Ontario and McMaster Osteoarthritis Index) Knee Stiffness Subscale Change From Baseline
Description: Knee stiffness assessment is made of 2 items; each has 5 possible values 0=none, 1=mild, 2=moderate, 3=severe, 4=extreme. The items are summed for a total range of 0 to 8. Therefore, the knee stiffness change from baseline range is -8 to 8. A negative change is a reduction in knee stiffness from the baseline knee stiffness score.
  A mixed-effect repeated measures regression model was used to estimate a least square mean for the entire "Measured Time Frame".
  Change from baseline was the dependent variable. Subject baseline score was a fixed effect covariate. Enrollment site, treatment, visit, and treatment by visit interaction were fixed class effects. Subject was a random effect. A least square mean single point estimate and 95%CI was calculated for the entire "Measured Time Frame" using all data collected at each time point within the "Measured Time Frame".
Time Frame: over 18 weeks (week timepoints 6, 10, 14, and 18)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | ARTZ | DUROLANE
Number analyzed (Participants) | 158 | 161
units on a scale | -1.73 [-1.87 to -1.59] | -1.87 [-2.00 to -1.73]
Statistical Analysis 1: Comparison: ARTZ vs DUROLANE; Ho: μDUR[18] - μArtz[18] ≥ +0.64 units Ha: μDUR[18] - μArtz[18] < +0.64 units; Test type: Non-Inferiority or Equivalence — This is a non-inferiority test. The non-inferiority margin of +0.64 units corresponds to an 8% margin on the knee stiffness subscale (range 0-8); Alpha inflation due to multiple testing was controlled using preplanned ordered stepwise hypothesis testing first over 18 weeks then over 26 weeks. This section reports the over 18 week knee stiffness subscale results; The eight and last step is to test Durolane WOMAC knee stiffness non-inferior to Artz WOMAC knee stiffness over 26 weeks; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.33 to 0.05]

8. Secondary Outcome: WOMAC (Western Ontario and McMaster Osteoarthritis Index) Knee Stiffness Subscale Change From Baseline
Description: as for outcome 7
Time Frame: over 26 weeks (week timepoints 6, 10, 14, 18, and 26)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | ARTZ | DUROLANE
Number analyzed (Participants) | 158 | 161
units on a scale | -1.80 [-1.93 to -1.67] | -1.95 [-2.08 to -1.82]
Statistical Analysis 1: Comparison: ARTZ vs DUROLANE; Ho: μDUR[26] - μArtz[26] ≥ +0.64 units Ha: μDUR[26] - μArtz[26] < +0.64 units; Test type: Non-Inferiority or Equivalence — This is a non-inferiority test. The non-inferiority margin of 0.64 units corresponds to an 8% margin on the knee stiffness subscale (range 0-8); Alpha inflation due to multiple testing was controlled using preplanned ordered stepwise hypothesis testing first over 18 weeks then over 26 weeks. This section reports the over 26 week knee stiffness subscale results; This is the eighth and last pre-planned hypothesis test; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-0.33 to 0.03]

ADVERSE EVENTS:
Time Frame: 26 weeks
Arm/Group | ARTZ | DUROLANE
Serious Adverse Events (participants affected / at risk) | 6/174 | 3/175
Other Adverse Events (participants affected / at risk) | 37/174 | 39/175
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ARTZ (N=174) | DUROLANE (N=175)
Coronary artery disease (Cardiac disorders) | 0 | 1
Otitis media (Ear and labyrinth disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Meniscus lesion (Musculoskeletal and connective tissue disorders) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 1
Colon polypectomy (Surgical and medical procedures) | 0 | 1
Cerebral infarction (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ARTZ (N=174) | DUROLANE (N=175)
Arthralgia (Musculoskeletal and connective tissue disorders) | 29 | 26
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 8 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No